CLINICAL TRIAL: NCT05461118
Title: Osteotomy Accuracy Using Mixed Reality Assisted Navigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Marshall Newman, Assistant Professor, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: [1829157
Record Dates: First submitted 2022-07-04; First posted 2022-07-15 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Osteotomy
Keywords: Mixed Reality Navigation

STUDY DESIGN:
Intervention Model Description: This is an interventional clinical trial, in which prospectively enrolled subjects will be compared with the historical control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Consented subjects will undergo osteotomies for their resective and reconstructive procedures using mixed reality adjuncts (Magic Leap ®, Microsoft Hololens ®) to commercially available navigation platforms (BrainLAB ®).
  Interventions: Procedure: Experimental:Treatment group

INTERVENTIONS:
Procedure: Experimental:Treatment group — Osteotomy surgical planning to be done using intraoperative mixed reality augmentation of a commercially available navigation platform.

SUMMARY:
An osteotomy is a standard surgical operation in which one or more bones are cut or lengthened or re-shaped. While planning for osteotomy, the surgeon sometimes uses a custom-manufactured cutting guide. The investigators are testing a relatively new approach called mixed reality navigation in planning this surgery in this study.

For the purpose of this study, the investigators will compare the accuracy of performing osteotomies with the aid of mixed reality navigation as compared to osteotomies that were performed using prefabricated cutting guides for patients in the past few years.

DETAILED DESCRIPTION:
The use of virtual surgical planning and custom cutting guide fabrication for craniomaxillofacial osteotomies is becoming more and more common, but it remains very expensive at present, particularly for cranial procedures. As such, many practitioners utilize open-source third-party software and in-house 3D printing to aid in reducing operating costs while maintaining surgical precision and accuracy as well as the benefits of decreased intraoperative time. The use of augmented and mixed reality platforms in craniomaxillofacial surgery has demonstrated usefulness in both preoperative planning and intraoperative visualization. It has been used in the past several years during craniofacial resective procedures, orthognathic surgery, dental implantology, and surgical education.

The purpose of investigating the accuracy of preplanned craniomaxillofacial osteotomies using the aid of a mixed reality platform viewer to augment currently available navigation platforms is to demonstrate a non-inferiority of the osteotomy technique compared to the current clinical gold standard for both precision and accuracy of craniomaxillofacial osteotomies - the use of custom patient-specific cutting guides based on preoperative virtual surgical planning.

The primary objective of this prospective study is to evaluate the accuracy of craniomaxillofacial osteotomies performed with the aid of mixed reality navigation as compared to osteotomies performed using prefabricated cutting guides for similar procedures that have been planned virtually preoperatively.

The secondary objective is to determine if osteotomies performed using mixed reality navigation can be effectively completed in a minimally invasive manner.

Hypothesis: Craniomaxillofacial osteotomies performed via the mixed reality navigation method can be completed with the same degree of accuracy to a preoperative virtual surgical plan as with the use of custom printed cutting guides or within 2 mm of variance.

Sample size: n=16 patients/group to achieve a power of 0.8 and a significance level of 0.05. The investigators expect to recruit 40 patients total for the study site, including a 20% drop rate for each group

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 16 years and older
* Has a benign or malignant mandibular or maxillary pathology who will require resection and who will undergo immediate reconstruction
* Consents to have resective and reconstructive procedures completed with the aid of mixed reality assisted navigation.

Exclusion Criteria:

1. Presence of acute infection at the time of surgery
2. Not able to speak in English or illiterate or lacking the decision-making capacity to consent for study.
3. Pregnant women because elective surgery is usually delayed until after delivery to avoid risks and complications associated with anesthetics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Measurements of osteotomy change on one-time post-operative imaging of CT scans | One time measurement completed within 1 month of surgery on postoperative CT scans of the face that are obtained within 3 weeks following surgery.
  3-dimensional depth mapping of postoperative CT scans overlaid on preoperative virtually planned osteotomy to assess for a change from the preoperative plan measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Marshall F Newman, DMD, Principal Investigator — Dental College of Georgia- Augusta University
Locations (1):
- Augusta University-Dental College of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be published in a peer-reviewed journal upon completion and presented at appropriate conferences.